CLINICAL TRIAL: NCT06370143
Title: Gastric Cancer Prevention: Understanding Precursor Lesions and Risk Factors for Progression to Cancer
Brief Title: A Study Collecting Health Information to Understand and Prevent Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 24-083
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Gastric Atrophy; Gastric Intestinal Metaplasia; Dysplasia; Gastric Adenocarcinoma; Gastric Cancer
Keywords: Gastric cancer; gastric adenocarcinoma; gastric atrophy; Gastric Intestinal Metaplasia; dysplasia; Memorial Sloan Kettering Cancer Center; 24-083
MeSH Terms: conditions — Gastritis, Atrophic; Stomach Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants with atrophic gastritis, intestinal metaplasia, and dysplasia: Participants with presence of atrophic gastritis, intestinal metaplasia, and dysplasia and risk of the progression of these lesions
  Interventions: Behavioral: Questionnaire
- Control Group: Healthy controls
  Interventions: Behavioral: Questionnaire
- Participants with gastric cancer: Participants with gastric cancer
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — The questionnaire on clinical, environmental, lifestyle, and dietary risk factors will be administered

SUMMARY:
The purpose of this study is to create a registry of participants with precursor lesions for gastric cancer, including gastric atrophy, intestinal metaplasia, and dysplasia. Normal controls and individuals with gastric cancer for comparison of baseline characteristics will also be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Able to read and understand English and Spanish
* Meet criteria for one of three potentially eligible study populations:

  * Individuals with gastric atrophy, gastric intestinal metaplasia, or dysplasia: Had a previous diagnosis of or have been diagnosed by the investigation team with gastric atrophy, gastric intestinal metaplasia, or dysplasia of the gastric mucosa on pathology review from an endoscopic biopsy. Individuals who have a prior history of early gastric cancer may be included, if they were treated endoscopically and have no evidence of disease. Individuals who have a prior history of a cancer other than upper gastrointestinal cancer may also be included, if they have no evidence of disease for at least 1 year prior to study enrollment and are not undergoing active treatment for any malignancy at any time throughout the study period
  * Healthy controls (average risk): Individuals with no history of cancer or gastric precursor lesions undergoing a clinically indicated endoscopy at MSK for workup or dyspepsia or reflux
  * Gastric cancer cases: Individuals with a known diagnosis of early gastric adenocarcinoma undergoing surgical resection at MSK

Exclusion Criteria:

* Age < 18 years old
* Women who are pregnant (may be enrolled after delivery)
* Individuals with a prior history of upper gastrointestinal surgery or a prior cancer who are undergoing active treatment for malignancy or have been diagnosed within 1 year prior to the study enrollment or with pancreatic cancer. (This does not include incidentally diagnosed primary gastric adenocarcinoma identified during study follow up. Individuals diagnosed with gastric carcinoid limited to the stomach will also be included, given their ongoing parallel risk for gastric adenocarcinoma.)
* Have severe comorbidities with expected survival time <2 years or which would prevent them from undergoing routine elective EGD (at the discretion of the patient's provider and the study team)
* Individuals having Hereditary Diffuse Gastric Cancer Syndrome, mutations including CDH1 and CTNNA1, or more than one genetic mutation
* Exclude high risk esophageal and duodenal lesions including:

  * Duodenal Adenoma
  * Dysplasia or cancer at the esophagus or gastroesophageal junction
* Patients with an increased risk for biopsies during EGD, such as those with clotting disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan Kettering (MSK).
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2036-04-11 (Estimated); Study Completion 2036-04-11 (Estimated)

PRIMARY OUTCOMES:
Creation of participant registry | Up to 10 years
  The primary objective of this study is to create a registry of individuals with precursor lesions for gastric cancer, including gastric atrophy, intestinal metaplasia, and dysplasia. Normal controls and individuals with gastric cancer for comparison of baseline characteristics will also be enrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Laszkowska, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org